CLINICAL TRIAL: NCT05071469
Title: Comparison of Short-term Effects of Two Different Treatment Methods in Patients With Subacromial Impingement Syndrome: a Randomized Controlled Single-blind Trial
Brief Title: Comparison of Two Different Treatment Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banu BAYAR (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Banu BAYAR, Principal investigator, Head of Physiotherapy and Rehabilitation Department, Pt. PhD. Prof., Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180030/16
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Subacromial Impingement Syndrome; Musculoskeletal Diseases; Musculoskeletal Injury; Musculoskeletal Pain; Weakness, Muscle
Keywords: Subacromial Impingement Syndrome; Mulligan Mobilization Technique; Kinesiotaping; Physiotherapy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Musculoskeletal Diseases; Musculoskeletal Pain; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (No Intervention): Control group
- Kinesiotaping Group (KG) (Experimental): Experimental group
  Interventions: Other: Kinesiotaping
- Mulligan Mobilization Technique Group (MG) (Experimental): Experimental group (2)
  Interventions: Other: Mulligan Mobilization Technique

INTERVENTIONS:
Other: Kinesiotaping — KT was applied.
  Arms: Kinesiotaping Group (KG)
Other: Mulligan Mobilization Technique — MMT was applied
  Arms: Mulligan Mobilization Technique Group (MG)

SUMMARY:
A number of previous studies investigated the effects of kinesiotaping (KT) in subacromial impingement syndrome (SIS).

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SIS) is characterized by shoulder pain that is exacerbated with especially arm elevation or overhead physical activities.

ELIGIBILITY:
Inclusion Criteria:

* Impingement symptoms in clinical tests
* Pain >1 month

Exclusion Criteria:

* Any shoulder pathology.
* Have chronic systemic diseases or infections.
* History of any surgery shoulder complex.
* steroid injections and therapeutic approaches

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change of pain severity | Baseline- after 2 weeks (after treatment)
  Via VAS.
Change of Range of Motion | Baseline- after 2 weeks (after treatment)
  Via goniometer.
Change of Functionality | Baseline- after 2 weeks (after treatment)
  Via SPADI.

SECONDARY OUTCOMES:
Change of Sleep Quality | Baseline- after 2 weeks (after treatment)
  Via VAS.
Change of Satisfaction of Life | Baseline- after 2 weeks (after treatment)
  Via SWLS.
Change of Satisfaction of Treatment | Baseline- after 2 weeks (after treatment)
  Via VAs.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided